CLINICAL TRIAL: NCT06541483
Title: A Multicenter Clinical Study of Ultra-Fast-Track Cardiac Anesthesia in Minimally Invasive Cardiac Surgery for Valvular Heart Disease
Brief Title: Multicentre Clinical Study of Ultra-Fast-Track Anaesthesia for Minimally Invasive Heart Valve Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); Fudan University (Other); Wuhan Asia Heart Hospital (Other); Tianjin Chest Hospital (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xiangya Hospital of Central South University (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 099
Record Dates: First submitted 2024-07-23; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Heart Valve Diseases; Enhanced Recovery After Surgery
Keywords: Ultra-fast-track Anesthesia; minimally invasive cardiac surgery
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-Fast-Track Cardiac Anesthesia(UFTCA) (Experimental): The researchers implemented an ultra-fast-track anesthesia protocol, and the tracheal tube was removed immediately or within 1 hour of awakening at the end of the operation.
  Interventions: Procedure: Ultra-Fast-Track Cardiac Anesthesia(UFTCA)
- conventional general anesthesia (CGA) (Other): The researcher implemented a conventional anesthesia protocol, and participants were not extubated at the end of the procedure and were admitted to the ICU under anesthesia with an endotracheal tube.
  Interventions: Procedure: conventional general anesthesia (CGA)

INTERVENTIONS:
Procedure: Ultra-Fast-Track Cardiac Anesthesia(UFTCA) — (UFTCA)The researcher removed the endotracheal tube either immediately or within 1 hour of the end of the procedure.
  Arms: Ultra-Fast-Track Cardiac Anesthesia(UFTCA)
Procedure: conventional general anesthesia (CGA) — (CGA)The researcher not extubated at the end of the operation and were admitted to the ICU under anesthesia with an endotracheal tube.
  Arms: conventional general anesthesia (CGA)

SUMMARY:
The goal of this clinical trial is to evaluate the clinical effects of ultra-fast-track anesthesia (UFTA) for minimally invasive cardiac surgery (MICS) in adults. It will also learn about the safety and feasibility of Ultra-Fast-Track cardiac surgery(UFTCA).The main questions it aims to answer are:Does UFTCA promote rapid postoperative recovery, reduce postoperative complications and perioperative mortality, and improve the quality of mid- and long-term survival.And does it improve patient satisfaction and reduce healthcare costs.

Participants will receive homogenized perioperative management in the cardiac ward, extracorporeal circulation, and postoperative ICU, except for anesthesia extubation time.Furthermore，Participants need complete quality of life scales at 30 days, 90 days, six months, and one year after surgery, separately.

Participants in this study are adults who required elective minimally invasive heart valve surgery under extracorporeal circulation.This study will be able to promote rapid recovery while reducing the associated costs and the financial burden on participants.Retrospective big data analysis of perioperative clinical characteristics of patients undergoing minimally invasive heart valve surgery to establish a risk warning model and develop a perioperative management program. The investigators then conducts a randomized group trial comparing the similarities and differences between conventional general anesthesia（CGA） and ultra-fast-track cardiac anesthesia(URTCA) to demonstrate the effectiveness and safety of UFTA in MICS.Finally, building expert consensus.

DETAILED DESCRIPTION:
This study was divided into two parts:The first part is retrospective data collection and organization, screening risk factors to establish an early warning model to improve the perioperative management program, and the other part is conducted using a randomized controlled trial to evaluate the effectiveness, safety and benefit of the perioperative management program of ultra-fast-track anesthesia(UFTA) for minimally invasive heart valve surgery. The specific program is as follows:

Part I

1. Establishment of an information collection platform Log in to the platform for electronic data entry and retain the paper version of the CaseReportForm（CRF）
2. Retrospective data collection Relying on the National Head Medical Center for Cardiac Surgery, 5000 perioperative case data of minimally invasive heart valve surgery patients were counted to obtain the perioperative clinical characteristics of Chinese adult minimally invasive heart valve surgery patients.
3. Screening for risk factors Statistical analysis of risk factors affecting perioperative ultra-fast-track anesthesia delivery and postoperative complications
4. Establishment of early warning model Combining age stratification, surgical mode stratification and general characteristics, establish an early warning model to improve the perioperative management protocol of ultra-fast channel anesthesia for minimally invasive heart valve surgery.

Part II Recruitment of participants for a prospective randomized controlled trial

1. Participants Patients undergoing elective minimally invasive adult heart valve surgery will be selected after completion of history taking, physical examination, preoperative laboratory and ancillary investigations, preoperative health and quality of life questionnaires, and frailty assessment of their physical condition, and will be confirmed to be free of any one of the "Exclusion Criteria" and to meet any one or more of the "Inclusion Criteria". Those who fulfill any one of the "Exclusion Criteria" and more than one of the "Inclusion Criteria" will be given a screening number. After completing the basic information and preoperative medications, the participant signed the informed consent form. If either the participant or the family member does not agree to participate in the study, the participant will only be given a screening number and the study will end here.
2. Randomized grouping Participants who were included to meet the criteria were randomly divided into the ultra-fast-track anesthesia group (UFTCA) and the conventional general anesthesia group (CGA), and the homogenized perioperative management of the extracardiac ward, extracorporeal circulation, and postoperative ICU was implemented, except for anesthesia resuscitation methods.
3. Anesthesia management 3.1 Preoperative Preoperative education, nutritional support, fasting and abstinence from food and drink, prophylactic multimodal analgesia (preoperative oral pregabalin 150 mg and acetaminophen 1000 mg) 3.2 Intraoperative Anesthesia mode: tracheal intubation general anesthesia plus nerve block anesthesia Induction of anesthesia: intravenous slow push etomidate fat milk injection 0.15 mg/kg, propofol injection 0.5~1.0 mg/kg, sufentanil citrate injection 0.4~0.5 mg/kg, rocuronium bromide 0.6~0.8 mg/kg, to be the patient's consciousness disappeared, to be the mask pressurized denitrification of oxygen for 3~5 minutes, muscle relaxation after the complete effect of the laryngoscopy under the direct visualization The patient was intubated, fixed, and mechanically ventilated, and the respiratory parameters were set as follows: Fraction of inspiratory oxygen concentration (FiO2): 50~80%, tidal volume (VT): 6~8 ml/kg, respiratory rate (RR): 10~12 times/min, Inhalation-exhalation ratio (I:E): 1:2, Maintain End-tidal CarbonDioxidePartialPressure (PetCO2) at 35~45 mmHg.

   Anesthesia maintenance: Propofol injection 150~250 μg/(kg·min) and remifentanil 0.2~0.4 μg/(kg·min) were continuously pumped through the central venous catheter, and intraoperative EEG Bispectral Index (BIS) values were maintained between 40~60.

   According to the hemodynamic indexes, respiratory parameters and the needs of surgical operation, intravenous sufentanil was injected in divided doses of 0.1~0.2 μg/kg, and the total amount of intraoperative sufentanil was controlled to be 1.0~1.5 μg/kg.

   Additional rocuronium bromide 0.1~0.2 mg/kg was added at the time of aortic blockade and opening, respectively.

   Intraoperative multimodal analgesia: (Pectoral nerves I(Pecs I), Pectoral nerves II(Pecs II), anterior serratus plane block(SPB)) anesthetic resuscitation: Evaluate to confirm whether the patient can be included in ultra-fast-track anesthesia.

   After the aorta was opened, the anesthesiologist, by observing the surgical procedure and communicating with the surgeon as well as the sonographer in a timely manner, confirmed that the surgery was successful, the heart was restarting normally, the extracorporeal circulation was withdrawn smoothly, there was no active hemorrhage in the surgical field, hemostasis was complete, oxygenation was functioning well, and the patient's finger pulse oximetry saturation was ≥98% under conditions of inhaled pure oxygen.

   UFTCA:The amount of propofol maintenance was dynamically adjusted according to the degree of stimulation at the beginning of chest closure, and all intravenous anesthesia maintenance drugs were discontinued at the beginning of chest closure. When the patient is under deep anesthesia, clear the patient's airway secretions and other foreign objects in advance; without interfering with the surgeon's operation, give bilateral lung bulging, and according to the trend of the BIS value and the patient's somatic reaction or not, give a single intravenous injection of propofol of 20~30mg as appropriate to maintain the patient's sedation until the end of the operation, and then remove the airway catheter when the patient is fully awake on the operating table. If necessary, an appropriate amount of neostigmine methylsulfate 1mg and atropine sulfate injection 0.5mg can be used intravenously to antagonize the muscle relaxant.

   CGA:Propofol injection 150~250 μg/(kg·min) and remifentanil 0.2~0.4 ug/(kg·min) were continuously pumped, and the patients were transferred to the ICU with tubes, and the ICU doctors decided the timing of stopping sedation and extubation.

   3.3 Postoperative multimodal analgesia Immediately after surgery, an intravenous analgesic pump was connected (sufentanil 200 μg and palonosetron 0.25 mg saline configured to a total of 200 mL)
4. Surgery Valve surgery encompasses aortic valve / mitral valve / tricuspid valve disease, performing single / double / triple valves, using minimally invasive procedures.This can be done through a small upper sternal incision, a small right anterior chest incision or a small transaxillary incision.
5. Extracorporeal circulation management The pre-filled fluid for extracorporeal circulation was 500~750 ml of crystalloid, 150 ml of 20% mannitol, 100 ml of 20% albumin, and 150 ml of sodium bicarbonate.

   Heparinization was performed at 3~4 mg/kg, and extracorporeal circulation was started after activated clotting time(ACT)>480s. The pacing fluid and dosage was 30 ml/kg, and the total amount did not exceed 2000 ml.

   During extracorporeal circulation, the mean arterial pressure was maintained at 50~80 mmHg, and the perfusion flow rate was 2.2~2.4 L/m^2.
6. Postoperative monitoring The Visual Analogue Score (VAS) was used for pain assessment after tracheal tube removal. VAS pain score by the nurse every 4 hours, if VAS ≥ 3, then press the analgesic pump once additional sufentanil 3 ~ 5 μg, 3 minutes later to assess again, if the patient VAS ≥ 3, then press the analgesic pump again additional sufentanil 3 ~ 5 μg; if sufentanil reached the analgesic pump set the limit of the amount of VAS ≥ 3 or produce serious nausea and vomiting and other side effects, then the intravenous oxycodone 10mg / time for Remedial analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤80 years
* American Society of Anaesthesiologists (ASA) class I-III
* New York Heart Association (NYHA) cardiac class III or below
* Preoperative inspired air pulse oximetry (SpO2) ≥95%
* Ejection fraction (EF) ≥ 40%
* No contraindications to nerve blocks

Exclusion Criteria:

* Patient's refusal to participate
* Severe communication disorders
* Severe disorders of coagulation with spontaneous bleeding tendency
* Long-term application of opioid analgesics
* Pulmonary hypertension (mean pulmonary artery pressure ≥55 mmHg)
* People who need artificial ventilation
* Allergy to dexmedetomidine and ropivacaine
* Complex aortic root surgery such as root widening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
tracheal tube extubation time | From the end of the operation to the removal of the tracheal tube,up to 3 days
  Time interval for tracheal extubation
ICU length of stay | From entry to exit from ICU,approximately 3 days
  Length of time participants stayed in the ICU
Post-operative hospitalization | From the end of surgery to discharge, approximately 1 week
  Length of postoperative hospitalization
Length of hospitalization | From admission to discharge, approximately 2 weeks
  Length of time participants stayed in the hospital
complication | From the end of surgery to 1 year after surgery
  Acute kidney injury, coma, acute respiratory distress syndrome (ARDS), postoperative atrial fibrillation, pericardial tamponade, gastrointestinal complications, death, cardiac arrest, heart block, and permanent stroke
Unscheduled events | From the end of surgery to 30 days after surgery
  reintubation, reoperation,ICU readmission, 30-day readmission
The 36-Item Short Form Health Survey(SF-36) | up to 1 year postoperative
  minimum values:0 maximum values:100 higher scores mean a better outcome
expenditure | From admission to discharge, approximately 2 weeks
  Total cost of treatment

SECONDARY OUTCOMES:
Time from end of surgery to removal from operating room | From end of surgery to removal from operating room, up to 1 hour
  Time from end of surgery to removal from operating room
Intraoperative opioid dosages | intraoperative
  Intraoperative dosage of sufentanil and remifentanil for induction and maintenance of anesthesia
VAS score | 72 hours post-surgery
  minimum values:1 maximum values:10 higher scores mean a worse outcome
Postoperative opioid dosage | From the end of surgery to discharge,approximately 1 week
  Level of postoperative analgesia
Application of vasoactive drugs | intraoperative
  Vasoactive drugs given as per participant and intraoperative needs
oxygenation index | From admission to discharge, approximately 2 weeks
  Pulmonary Function Assessment
Thoracic drainage within 24 hours | 24 hours post-surgery
  Thoracic drainage within 24 hours after surgery
Total Thoracic Drainage | From the end of surgery to chest drain removal, approximately 3 days
  Total postoperative chest drainage
Thoracic drain removal time | From the end of surgery to chest drain removal, approximately 3 days
  Thoracic drain removal time
Bowel evacuation time | Time from end of surgery to first bowel evacuation, approximately 2 days
  Assessment of postoperative recovery of gastrointestinal function
time out of bed | Time from end of surgery to first time out of bed, approximately 2 days
  First time out of bed
Inflammatory levels | From the start of anesthesia induction to 48 hours after extubation
  interleukin(IL)-1β,IL-4,IL-6,IL-8,IL-10,Procalcitonin(PCT),Hypersensitive C-reactive protein(hs-CRP) and tumor necrosis factor(TNF)-α
coagulation | One day before to the next day after surgery,72 hours
  Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR), Fibrinogen (FIB), D-dimer (DD2), Fibrin (Pro) Degradation Product (FDP), Antithrombin III (ATIII ), Thromboelastography (TEG)
myocardial injury | One day before to the next day after surgery,72 hours
  N-terminal Pro-brain B-type Natriuretic Peptides(NT-proBNP）, Cardiac troponin I(cTnI )
neurological injury | One day before to the next day after surgery,72 hours
  Neuron-specific enolase(NSE)
Anesthesia costs | Until 1 hours post-surgery
  Costs incurred for perioperative anesthesia medications and anesthesia management requirements
Patient satisfaction | up to 1 year after discharge from hospital
  Participants are rated on a 10-point satisfaction scale minimum values:1 maximum values:10 higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mei J Yan, QC, Study Chair — Zhejiang Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krzych L, Kucewicz-Czech E. It is time for enhanced recovery after surgery in cardiac surgery. Kardiol Pol. 2017;75(5):415-420. doi: 10.5603/KP.a2017.0014. Epub 2017 Feb 2. No abstract available. PMID 28150277
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Coleman SR, Chen M, Patel S, Yan H, Kaye AD, Zebrower M, Gayle JA, Liu H, Urman RD. Enhanced Recovery Pathways for Cardiac Surgery. Curr Pain Headache Rep. 2019 Mar 14;23(4):28. doi: 10.1007/s11916-019-0764-2. PMID 30868281
- [Background] Zaouter C, Imbault J, Labrousse L, Abdelmoumen Y, Coiffic A, Colonna G, Jansens JL, Ouattara A. Association of Robotic Totally Endoscopic Coronary Artery Bypass Graft Surgery Associated With a Preliminary Cardiac Enhanced Recovery After Surgery Program: A Retrospective Analysis. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):1489-97. doi: 10.1053/j.jvca.2015.03.003. Epub 2015 Mar 5. PMID 26119408
- [Background] Fleming IO, Garratt C, Guha R, Desai J, Chaubey S, Wang Y, Leonard S, Kunst G. Aggregation of Marginal Gains in Cardiac Surgery: Feasibility of a Perioperative Care Bundle for Enhanced Recovery in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):665-70. doi: 10.1053/j.jvca.2016.01.017. Epub 2016 Jan 16. PMID 27321791
- [Background] Williams JB, McConnell G, Allender JE, Woltz P, Kane K, Smith PK, Engelman DT, Bradford WT. One-year results from the first US-based enhanced recovery after cardiac surgery (ERAS Cardiac) program. J Thorac Cardiovasc Surg. 2019 May;157(5):1881-1888. doi: 10.1016/j.jtcvs.2018.10.164. Epub 2018 Dec 8. PMID 30665758
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Pokhrel S, Gregory A, Mellor A. Perioperative care in cardiac surgery. BJA Educ. 2021 Oct;21(10):396-402. doi: 10.1016/j.bjae.2021.05.008. Epub 2021 Jul 13. No abstract available. PMID 34567795
- [Background] Cohen B, Turan A. Enhanced recovery after cardiac surgery - Is evidence still necessary? J Clin Anesth. 2019 May;54:171-172. doi: 10.1016/j.jclinane.2018.12.049. Epub 2018 Dec 29. No abstract available. PMID 30599274
- [Background] Noss C, Prusinkiewicz C, Nelson G, Patel PA, Augoustides JG, Gregory AJ. Enhanced Recovery for Cardiac Surgery. J Cardiothorac Vasc Anesth. 2018 Dec;32(6):2760-2770. doi: 10.1053/j.jvca.2018.01.045. Epub 2018 Jan 31. PMID 29503121
- [Background] Bianchi P, Constantine A, Costola G, Mele S, Shore D, Dimopoulos K, Aw TC. Ultra-Fast-Track Extubation in Adult Congenital Heart Surgery. J Am Heart Assoc. 2021 Jun;10(11):e020201. doi: 10.1161/JAHA.120.020201. Epub 2021 May 17. PMID 33998289
- [Background] Zayat R, Menon AK, Goetzenich A, Schaelte G, Autschbach R, Stoppe C, Simon TP, Tewarie L, Moza A. Benefits of ultra-fast-track anesthesia in left ventricular assist device implantation: a retrospective, propensity score matched cohort study of a four-year single center experience. J Cardiothorac Surg. 2017 Feb 8;12(1):10. doi: 10.1186/s13019-017-0573-9. PMID 28179009
- [Background] Xu J, Zhou G, Li Y, Li N. Benefits of ultra-fast-track anesthesia for children with congenital heart disease undergoing cardiac surgery. BMC Pediatr. 2019 Dec 11;19(1):487. doi: 10.1186/s12887-019-1832-9. PMID 31829170
- [Background] Akhtar MI, Momeni M, Szekely A, Hamid M, El Tahan MR, Rex S. Multicenter International Survey on the Clinical Practice of Ultra-Fast-Track Anesthesia with On-Table Extubation in Pediatric Congenital Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):406-415. doi: 10.1053/j.jvca.2018.07.006. Epub 2018 Jul 7. PMID 30115517
- [Background] Jiang S, Wang L, Teng H, Lou X, Wei H, Yan M. The Clinical Application of Ultra-Fast-Track Cardiac Anesthesia in Right-Thoracoscopic Minimally Invasive Cardiac Surgery: A Retrospective Observational Study. J Cardiothorac Vasc Anesth. 2023 May;37(5):700-706. doi: 10.1053/j.jvca.2023.01.010. Epub 2023 Jan 13. PMID 36804223
- [Background] Ahmad U, Khattab MA, Schaelte G, Goetzenich A, Foldenauer AC, Moza A, Tewarie L, Stoppe C, Autschbach R, Schnoering H, Zayat R. Combining Minimally Invasive Surgery With Ultra-Fast-Track Anesthesia in HeartMate 3 Patients: A Pilot Study. Circ Heart Fail. 2022 May;15(5):e008358. doi: 10.1161/CIRCHEARTFAILURE.121.008358. Epub 2022 Mar 7. PMID 35249368
- [Background] Feng J, Wang H, Peng L, Xu H, Song X. Effects of Thoracic Paravertebral Block on Postoperative Analgesia in Infants and Small Children undergoing Ultra-Fast Track Cardiac Anesthesia: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2023 Apr;37(4):539-546. doi: 10.1053/j.jvca.2022.12.006. Epub 2022 Dec 11. PMID 36717316